CLINICAL TRIAL: NCT00561613
Title: A Phase I Postcoital Testing and Safety Study of the SILCS Diaphragm, Prototype VI
Brief Title: Postcoital Testing of the SILCS Diaphragm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Jill Schwartz, MD/Project Leader, CONRAD
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A02-081
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Contraceptive Device
Keywords: Diaphragm; postcoital test; SILCS; nonoxynol-9
MeSH Terms: interventions — Lubricants; Spermatocidal Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): SILCS with K-Y Jelly
  Interventions: Other: SILCS and lubricant
- 2 (Active Comparator): SILCS with N-9
  Interventions: Other: SILCS and spermicide

INTERVENTIONS:
Other: SILCS and lubricant
  Arms: 1
Other: SILCS and spermicide
  Arms: 2

SUMMARY:
This was a Phase I multi-center, randomized study in 40 healthy, sexually active women not at risk for pregnancy due to previous female sterilization. The male partners of the participants were consented to participate in the study. The clinician evaluating the cervical mucus for midcycle characteristics and presence of sperm was blinded as to gel used. The product tested was the SILCS diaphragm with Gynol II (spermicide) and the SILCS diaphragm with KY Jelly (lubricant). The sequence of diaphragm and gel use was determined by randomization. The study was conducted at two centers, Magee-Womens Hospital in Pittsburgh, Pennsylvania and CONRAD's Clinical Research Center at the Eastern Virginia Medical School in Norfolk, Virginia.

The study consisted of a screening visit, a baseline cycle, and up to 2 cycles of post-coital tests (PCTs) for a total of 7 visits. The first PCT was a baseline PCT, performed without the use of any product, in order to demonstrate the subject's ability to produce receptive, midcycle cervical mucus. The partner's ability to produce motile sperm capable of penetrating the cervical mucus was evaluated in this cycle. Test PCTs were carried out during the second and third menstrual cycle using either the SILCS diaphragm with N-9 or the SILCS diaphragm with lubricant. Cycles were repeated depending on the characteristics of the cervical mucus and the number of sperm found in the vaginal pool and endocervical specimens; thus, some women may undergo more than three PCTs. An additional test cycle with a modified polymer spring device was performed in a subset of participants.

Colposcopy was performed during the mucus check and post-coital test visits in all three cycles in order to document the baseline condition of the vagina and cervix pre- and post-intercourse and, in test cycles, to note the effect of product.

Vaginal samples were taken from the posterior fornix of the vagina and the cervical os at each visit during the baseline and test cycles to measure for the presence of PSA.

ELIGIBILITY:
Inclusion Criteria:

1. Female Participants

   * 18-45 years old (inclusive)
   * In good general health based on medical history & physical exam
   * Previous bilateral tubal ligation or salpingectomy
   * Regular menstrual cycles of 24-35 days (inclusive)
   * Negative urine pregnancy test at admission
   * Not currently breast feeding
   * No significant gynecological abnormalities
   * Normal cervical Papanicolaou smear within 6 months preceding enrollment
   * In a stable relationship with only one sexual partner
   * Willing to undergo at least three PCTs
   * Willing to abstain from intercourse and use of vaginal products
   * Willing to use condoms from day 1 of each menstrual cycle until midcycle
2. Male Participants

   * Age 18 years and older
   * Able and willing to provide written informed consent
   * Willing to engage in intercourse with and without condoms

Exclusion Criteria:

1. Female Participants

   * History in subject of allergy to study products
   * Positive wet mount for Trichomonas vaginalis
   * History of any STD within 6 months of enrollment
   * Device does not appropriately fit volunteer, as determined by clinician
   * Inability to insert, position, and/or remove study device
   * Participation in another study within 30 days prior to enrollment
2. Male Participants

   * History of allergy to study products
   * History of vasectomy
   * In the six months prior to study, diagnosed with or treated for any STI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2003-08; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Percentage of women with any sperm in the cervical mucus, with ≥ 5 progressively motile sperm per high power field (HPF), and the average number of progressively motile sperm per HPF. | Within 2-3 hours of intercourse.

SECONDARY OUTCOMES:
Symptoms and signs of irritation of the external genitalia, cervix, and vagina before and after intercourse and by gel product. The handling, fit, and general acceptability of the SILCS diaphragm was assessed. | Before and after intercourse

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, MD, Study Director — CONRAD
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Derived] Schwartz JL, Ballagh SA, Creinin MD, Rountree RW, Kilbourne-Brook M, Mauck CK, Callahan MM. SILCS diaphragm: postcoital testing of a new single-size contraceptive device. Contraception. 2008 Sep;78(3):237-44. doi: 10.1016/j.contraception.2008.04.118. Epub 2008 Jul 3. PMID 18692615